CLINICAL TRIAL: NCT00328315
Title: Myocardial Perfusion SPECT Using a Rotating Multi-segment Slant-hole Collimator
Brief Title: Cardiac SPECT With Rotating Slant Hole Collimator
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: NO:05-06-03-02; R01 EB 0019-83 (Other: NIH)
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Diseases; Chest Pain
Keywords: Myocardial Perfusion SPECT
MeSH Terms: conditions — Coronary Artery Disease; Chest Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
The goal is to conduct a clinical pilot study to evaluate the use of a rotating multi-segment slant-hole collimator in the detection of myocardial defects.

DETAILED DESCRIPTION:
Myocardial perfusion SPECT is recognized as an effective clinical diagnostic imaging technique in the assessment of myocardial perfusion and coronary artery diseases. It is the most important clinical application of SPECT imaging techniques.

The goal is to conduct a clinical pilot study to evaluate the use of rotating multi-segment slant-hole (RMSSH) SPECT in the detection of myocardial defects especially in very sick patients in the nuclear medicine clinics, emergence room, and intensive care units. Comparison of the clinical utilities of the cardiac RMSSH SPECT technique with conventional cardiac planar and SPECT with parallel-hole collimation will also allow us to evaluate the potential application of the technique to a wider patient population.

The objective of this study is to test the hypothesis that quantitative 99mTc myocardial perfusion RMSSH SPECT provides similar diagnostic accuracy in patients with cardiac diseases as conventional SPECT imaging techniques.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 18-80 who are scheduled for a clinical Cardiac Stress Test

Exclusion Criteria:

* Pregnant Women and Children

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and Females 18-80 who are scheduled for a clinical Cardiac Stress Test
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Tsui, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States